CLINICAL TRIAL: NCT06888388
Title: Long-term Oncologic Safety of Nipple Sparing Mastectomy in Women With High Penetrance Germline Pathogenic Variants in Breast Cancer Susceptibility Genes
Brief Title: Long-term Safety of Nipple Sparing Mastectomy in Women With High Penetrance Breast Cancer Susceptibility Genes in Breast Cancer
Acronym: NSM
Status: Recruiting | Type: Observational
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Collaborators: Cancer Research Society (Other); Quebec Breast Cancer Foundation (Other)
Responsible Party: Principal Investigator, Stephanie Wong, Assistant Professor of Surgery, Sir Mortimer B. Davis - Jewish General Hospital
Other Study IDs: MP-05-2025-4291 (MP)
Record Dates: First submitted 2025-03-15; First posted 2025-03-21 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer Surgery
Keywords: breast cancer surgery; nipple sparing mastectomy; oncologic safety; Cancer prevention; Breast Cancer Prevention; BRCA; germline pathogenic variant; GPV; Li Fraumeni; Hereditary lobular breast cancer; Cowden syndrome; PALB2
MeSH Terms: conditions — Li-Fraumeni Syndrome; Hamartoma Syndrome, Multiple | interventions — Mastectomy, Subcutaneous; Mastectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Risk Reducing Mastectomy
  Interventions: Procedure: Nipple Sparing Mastectomy (NSM); Procedure: Skin-Sparing Mastectomy (SSM); Procedure: Total (Simple) Mastectomy
- Active surveillance

INTERVENTIONS:
Procedure: Nipple Sparing Mastectomy (NSM) — Nipple sparing mastectomy (NSM) is a surgical procedure which removes all macroscopic breast glandular tissue while retaining the skin as well as the nipple areola complex.
  Groups: Risk Reducing Mastectomy
Procedure: Skin-Sparing Mastectomy (SSM) — Skin sparing mastectomy (SSM) is a procedure that removes the nipple and areola complex along with all visible macroscopic breast glandular tissue.
  Groups: Risk Reducing Mastectomy
Procedure: Total (Simple) Mastectomy — Total (Simple) Mastectomy is a traditional mastectomy approach that removes the breast glandular tissue with a large overlying area of skin including the nipple and areola complex to allow for flat closure.
  Groups: Risk Reducing Mastectomy

SUMMARY:
Patients with a germline pathogenic variant (GPV) in high-penetrance breast cancer susceptibility genes who are considering risk reducing mastectomy (RRM) often strongly desire to keep their nipple areola complex but inquire as to whether it is safe to do so. Relative to traditional or skin sparing mastectomy (SSM) techniques, nipple sparing mastectomy (NSM) is associated with improved psychosocial and sexual well-being and is significantly better for body image and reducing feelings of disfigurement.

Despite this, guidelines have yet to endorse the use of NSM over other RRM techniques, stating that more data and longer follow-up are needed to confirm it as a safe and effective strategy in GPV carriers. As NSM was not routinely adopted in high-risk patient populations undergoing RRM before 2010, there has been little data to inform the long-term oncologic safety of NSM. Well-designed studies have reported low to negligible rates of subsequent breast cancer in BRCA1/2 carriers following NSM, but have been limited by short median follow-up of less than 3 years. The current study is designed to confirm, with longer follow-up, prior findings on the oncologic safety of NSM in unaffected BRCA1/2 carriers. The investigators will also expand data to other high-penetrance GPV carriers, including PALB2, CDH1, PTEN, and TP53, for whom there is little-to-no data on outcomes following RRM.

ELIGIBILITY:
Inclusion Criteria:

* Assigned female sex at birth
* Age 18 years or older
* Confirmed GPV in BRCA1, BRCA2, PALB2, TP53, CDH1 or PTEN identified on pre-symptomatic genetic testing

Exclusion Criteria:

* History of breast cancer prior to genetic testing
* History of ovarian cancer prior to genetic testing
* History of bilateral mastectomy performed prior to genetic testing
* Presence of a variant of uncertain significance (VUS) in the absence of another GPV in BRCA1, BRCA2, PALB2, TP53, CDH1 or PTEN.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Female patients aged 18-years or older with a confirmed GPV in BRCA1, BRCA2, PALB2, TP53, CDH1 or PTEN identified on pre-symptomatic genetic testing performed between January 1, 1994-June 30, 2024
Sampling Method: Non-Probability Sample
Enrollment: 4700 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of breast cancer following RRM | 10 years
  The primary outcome of interest is the incidence of breast cancer following RRM, defined as a histologically confirmed diagnosis of in situ or invasive breast cancer present within the nipple/areola, skin, subcutaneous tissue of the chest wall/reconstructed breast, or axillary lymph nodes. Patients with clinically occult invasive breast cancer diagnosed at the time of RRM (ie. on mastectomy pathology) will be excluded from the primary outcome analysis.

SECONDARY OUTCOMES:
Incidence of RRM | 10 years
  To evaluate uptake of RRM versus active surveillance amongst an international cohort of unaffected women with high-penetrance GPVs in BRCA1/2, PALB2, CDH1, PTEN, or TP53
Incidence of post-operative complications | 10 years
  To evaluate post-operative complications and supplemental surgery following NSM, SSM, and total mastectomy in those undergoing RRM
Incidence of pathologic outcomes following NSM | 10 years
  To evaluate pathologic outcomes following RRM, including the presence of high-risk lesions or occult in situ and/or invasive malignancy
Number of participants using endocrine prevention | 10 years
  To explore the use of endocrine prevention in unaffected women with high-penetrance GPVs in BRCA1/2, PALB2, CDH1, PTEN, or TP53 who elect to undergo active surveillance
Number of participants who have undergone pre-mastectomy imaging and post-mastectomy surveillance | 10 years
  To assess practices in pre-mastectomy imaging and post-mastectomy surveillance, including the number of participants who underwent preoperative MRI and mammography as well as post-mastectomy surveillance, including MRI, ultrasound and chest wall examination.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (4):
  - Yale University, New Haven, Connecticut
  - Brigham and Women's Hospital - Dana-Farber Brigham Cancer Center, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center (MSKCC), New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
- University of Melbourne, Peter MacCallum Cancer Center, Melbourne, Australia
- Ziekenhuis Aan de Stroom, Antwerp, Belgium
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - Hamilton Health Sciences, Hamilton, Ontario
  - Women's College Hospital, University of Toronto, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Quebec Université laval, Québec, Quebec
- Champalimaud Foundation, University of Lisbon, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No